CLINICAL TRIAL: NCT01123057
Title: Riboflavin-UVA Induced Collagen Crosslinking Treatment for Corneal Ectasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Lim Li, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R573/61/2007
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Corneal Ectasia
Keywords: keratoconus; collagen cross-linking; LASIK ectasia; keratoconus,lasik ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: riboflavin-induced collagen cross-linking treatment — The principle of the procedure is to induce collagen crosslinking of the corneal stroma by the using riboflavin/UVA-treatment.
  The technique involves topical application of riboflavin/dextran solution onto eye after removal of corneal epithelium. After initial riboflavin application for 30 minutes, UVA light is shone onto the cornea for another 30 minutes with continued topical riboflavin application.
Device: Riboflavin-UVA induced collagen cross-linking treatment for corneal ectasia — Use of riboflavin eyedrops during the procedure Use of UVA device (Peschke Meditrade)

SUMMARY:
This is a hospital-based interventional prospective study. Patients with clinical keratoconus or LASIK keratectasia presenting to the Singapore National Eye Centre who meet the eligibility criteria are recruited for this study. The aim of the study is to assess the safety and efficacy of riboflavin-UVA induced cross-linking treatment for corneal ectasia

DETAILED DESCRIPTION:
The purpose of this evaluation is to assess the safety and efficacy of riboflavin-UVA induced cross-linking treatment for corneal ectasia due to keratoconus and LASIK keratectasia. The principle of the procedure is to induce collagen crosslinking of the corneal stroma by the using riboflavin/UVA-treatment.

The technique involves topical application of riboflavin/dextran solution onto eye after removal of corneal epithelium. After initial riboflavin application for 30 minutes, UVA light is shone onto the cornea for another 30 minutes with continued topical riboflavin application.

A thorough examination is performed to evaluate the following pre-operatively:

* Manifest refraction results - Uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA)
* Cycloplegic refraction results - Uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA)
* Slit-lamp biomicroscopy and photography
* Intraocular pressure measurement
* Fundoscopy
* Corneal topography using Orbscan II and Pentacam
* Corneal aberrometry measurement using Technolas Zywave Aberrometer
* Endothelial cell count measurement using Konan noncontact endothelial cell analyser
* Confocal microscopy
* Corneal hysteresis measurement using Ocular Response Analyser
* Subjective feedback about quality of vision (VF 14 assessment) Post-operative Assessment (1 day, 1 week, 1 month, 3 months, 6 months and 1 year postoperatively)
* Uncorrected visual acuity and best corrected visual acuity with manifest refraction
* Cycloplegic refraction results - uncorrected visual acuity and best corrected visual acuity
* Subjective visual outcome rating
* Slit lamp examination and photography
* Fundoscopy
* Corneal topography
* Aberrometry measurement
* Endothelial cell count
* Confocal microscopy
* Corneal hysteresis measurement
* Report adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinical evidence of keratoconus or LASIK keratectasia (moderate to severe)
* Visual acuity with contact lenses must be better than or equal to 6/12 (20/40).
* Patients must be intolerant of contact lenses, i.e., they must be unable to wear contact lenses for a whole day.
* Patients should have a minimum of corneal thickness of 400um (with cornea at swollen state denuded of epithelium during surgery).
* In terms of general health, patients must not have any illnesses posing an immediate threat to life.
* Patients must over 18 years of age.
* Patients' contact lens wear must be stopped 3 days prior to preop assessment
* Patients can wear their lenses up to the day before the surgery
* Any vitamin C intake must be stopped 1 week prior to surgery
* Both eyes may be recruited if eligible.
* Patients with other non-inflammatory corneal thinning disorders such as pellucid marginal degeneration, keratoglobus and posterior keratoconus may be recruited

Exclusion Criteria:

* corneal thickness <400 µm in swollen state
* epithelial healing disorders (e.g. map-dot-fingerprint dystrophy, rheumatic disorders)
* refractive keratotomies
* corneal melting conditions
* herpes keratitis (UV can activate this herpes virus)
* associated systemic disorder such as Down's syndrome
* Pregnancy
* Breast-feeding.
* Patients with history of herpetic keratitis.
* Patients with autoimmune diseases
* Patients with IOP >21mmHg
* Patients with cataracts
* Patients taking part in other biomedical research in the 30 days prior to the start of this study.
* Patients with alcohol abuse, psychological weakness, or an uncooperative disposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
corneal topography | 1 year
  The keratometry values will be monitored.

SECONDARY OUTCOMES:
visual acuity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Li Lim, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T. Long-term results of riboflavin ultraviolet a corneal collagen cross-linking for keratoconus in Italy: the Siena eye cross study. Am J Ophthalmol. 2010 Apr;149(4):585-93. doi: 10.1016/j.ajo.2009.10.021. Epub 2010 Feb 6. PMID 20138607